CLINICAL TRIAL: NCT04583878
Title: FUVID Study: A Multi-center, Prospective Study Evaluating Exercise Intolerance and Dyspnea on Exertion in Patients Following First-episode Deep Venous Thrombosis and Pulmonary Embolism
Brief Title: FUVID Study: Functional Characterization of Children With Chronic Venous Thromboembolic Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ayesha Zia, Associate Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-0868
Record Dates: First submitted 2020-09-22; First posted 2020-10-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research Biomarkers: blood for inflammatory markers, thrombin generation and fibrinolysis assays are required for all participants. Research Blood for DNA/RNA only collected for those participants who consent to genetic material.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Pulmonary Embolism: The target accrual is based on the primary endpoint (exercise intolerance and dyspnea on exertion). To achieve adequate power and precision in the primary analysis, the target enrollment is 80 children. Both males and females of all races and ethnic groups are eligible for this study.
  Interventions: Diagnostic Test: Blood draw (Visit 1); Diagnostic Test: Blood draw (Visits 2 and 3)
- Control Group: A positive control group that has not had pulmonary embolism (PE) but is prescribed physical activity restrictions expected to produce a similar deconditioning effect as patients with PE will be enrolled from UT Southwestern only (cohort 1) or children who are no prescribed physical activity restrictions and are otherwise considered healthy (cohort 2). The target accrual of the positive control group is based on feasibility and availability of funds and will be limited to 25 controls.
  Interventions: Diagnostic Test: Blood draw (Visits 2 and 3)

INTERVENTIONS:
Diagnostic Test: Blood draw (Visit 1) — Labs will be drawn at Visit 1, also referred to as screening (within 60 days of diagnosis) with the standard of care labs drawn.
  Groups: Participants with Pulmonary Embolism
Diagnostic Test: Blood draw (Visits 2 and 3) — Labs will be drawn at Visit 2 (12 weeks post-diagnosis with a range of 10-16 weeks) and Visit 3 (12 months ± 30 days) for research purposes only and will be collected at Children's Medical Center and processed at UT Southwestern Medical Center.

SUMMARY:
This is a multi-center prospective cohort study of patients with first-episode deep venous thrombosis and pulmonary embolism.

DETAILED DESCRIPTION:
Subjects will be identified from the clinical setting and approached to participate in this observational study where participants will be enrolled at 3 different sites and referred from several more sites and have: cardiopulmonary exercise testing and pulmonary function testing at The Institute of Exercise and Environmental Medicine (IEEM), UTSW Exercise Facility, Cardiac MRI and MRI for pulmonary perfusion at Children's Medical Center and MR Spectroscopy and MR for Muscle Perfusion at the Advanced Imaging Research Center (AIRC) performed in Dallas over a 3 day research visit at week 12 and Month 12. Blood is collected for biomarkers at these visits and multiple questionnaires are completed by participants.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 to ≤ 21 years
* Participant must be able to speak and understand English
* Be willing to participate and able to comply with the study protocol
* For participants with PE: Children with acute, radiologically confirmed pulmonary embolism (PE) with our without DVT
* For control group: Cohort 1: Children who are prescribed physical activity restrictions for 2 up to 12 weeks following any minor outpatient surgery or, minor injury (surgery or injury is referred to as "diagnosis" hereafter) Cohort 2: Children who are not prescribed physical activity restrictions and are otherwise considered to be healthy.

Exclusion Criteria:

* Congenital heart disease with abnormal pulmonary circulation or with in-situ pulmonary artery thrombosis
* Chronic kidney disease
* Chronic inflammatory or an autoimmune disorder (such as systemic lupus erythematosus, juvenile rheumatoid disorder, inflammatory bowel disease, and sickle cell disease)
* A metabolic or endocrinological disorder such as diabetes mellitus or thyroid disorder
* History of or active cancer
* Pregnant
* Musculoskeletal limitations to exercise expected to be present uptil 4 months post-diagnosis
* Weight ≥ 300 lbs
* Contraindications to magnetic resonance imaging
* Frequent severe exacerbations of asthma defined by two or more bursts of systemic glucocorticoids (more than three days each) in the previous year or at least one hospitalization, intensive care unit stay or mechanical ventilation in the previous year. Patients should also be excluded if there are daily symptoms of asthma requiring daily use of short-acting bronchodilators such as albuterol or levalbuterol administration. The use of controller medications such as daily inhaled corticosteroids for mild persistent asthma is not exclusionary.
* Has any other medical condition, which in the opinion of the investigator may potentially compromise the safety or compliance of the patient or may preclude the patient's successful completion of the clinical study

Additional exclusion criteria for participants with PE:

* Prior history of DVT or PE (upper extremity, cerebral sinus venous thrombosis and abdominal thromboses encountered as a neonate are not exclusion criteria)
* Lack of anticoagulant treatment for the acute VTE due to contraindications

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will include children (defined as persons who have not attained the legal age for consent to treatments or procedures involved in the research, under the applicable law of the jurisdiction in which the research will be conducted), and patients (defined as individuals in a clinical setting with whom there is a treatment relationship).
  Participants must meet the eligibility criteria in order to participate in this trial.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in exercise capacity | 3 months and 12 months post-diagnosis
  Measured objectively by peak oxygen uptake (VO2) as a percent predicted based on ml/min/kg of lean body mass during cardiopulmonary exercise testing (CPET)
Change in dyspnea on exertion (DOE) | 3 months and 12 months post-diagnosis
  measured using Borg questionnaire and defined as a mean difference of > 1 between those with and without exercise intolerance at the end of the warm-up and submaximal work rates during CPET

SECONDARY OUTCOMES:
Change in cardiac maladaptation | 3 months and 12 months post-diagnosis
  Measured as ventriculo-arterial coupling ratio in response to exercise (change in Ea/Emax from rest to peak intensity exercise) during exercise cardiac magnetic resonance imaging (MRI)
Change in pulmonary/ventilatory limitations | 3 months and 12 months post-diagnosis
  Measured as VE/VCO2 in participants with and without exercise intolerance during cardiopulmonary testing
Change in muscle metabolic aberrations | 3 months and 12 months post-diagnosis
  Measured by % phosphocreatine (PCr) depletion (Δ %PCr) during exercise using 31P magnetic resonance spectroscopy on 7 Tesla in participants with and without exercise intolerance
Change in pulmonary vascular obstruction score in participants with and without exercise intolerance (Quantitative assessment) | At diagnosis, 3 months and 12 months post-diagnosis
  Quantitative Assessment: Measured using Qanadli Index scale (range 0-40; 0=minimum score and 40=maximum score) at pulmonary embolism diagnosis and 3 months post-diagnosis.
Change in pulmonary vascular obstruction score in participants with and without exercise intolerance (Qualitative assessment) | At diagnosis, 3 months and 12 months post-diagnosis
  Qualitative Assessment: Measured using pulmonary perfusion maps at diagnosis, 3 and 12 months post-diagnosis. Since qualitative, there are no minimum or maximum values.
Change in calf muscle perfusion and venous flow in participants with and without exercise intolerance and between affected and non-affected extremity | 3 months and 12 months post-diagnosis
  Measured using extremity arterial spin labelling on 7 Tesla MRI
Change in dyspnea ratings using Dalhousie Pictorial Scale | 3 months and 12 months post-diagnosis
  Measured at rest, fatigue, and post-exercise in participants with and without exercise intolerance
  Dalhousie Pictorial Scale measuring Dyspnea and Perceived Exertion (minimum score=4; maximum score=28; higher score means worse dyspnea)
Change in dyspnea ratings using Borg Dyspnea Scale | 3 months and 12 months post-diagnosis
  Measured at rest, fatigue, and post-exercise in participants with and without exercise intolerance
  Borg Dyspnea Scale (minimum score=0; maximum score=10; higher score means worse dyspnea)
Change in dyspnea ratings using Dyspnoea-12 Scale | 3 months and 12 months post-diagnosis
  Measured at rest, fatigue, and post-exercise in participants with and without exercise intolerance
  Dyspnoea-12 Scale (minimum score=0; maximum score=36; higher score means worse dyspnea)
Change in dyspnea ratings using Modified Medical Research Council Dyspnea Scale | 3 months and 12 months post-diagnosis
  Measured at rest, fatigue, and post-exercise in participants with and without exercise intolerance
  Modified Medical Research Council Dyspnea Scale (minimum score=0; maximum score=4; higher score means worse dyspnea)
Change in inflammatory cytokine biomarker - High-sensitivity CRP | At diagnosis, 3 months and 12 months post-diagnosis
  Measure inflammatory cytokine biomarker high-sensitivity CRP (unit of measure: mg/L) in participants with and without exercise intolerance
Change in inflammatory cytokine biomarkers - IL-6 and TNF | At diagnosis, 3 months and 12 months post-diagnosis
  Measure inflammatory cytokine biomarkers IL-6 and TNF-α (unit of measure: pg/mL) in participants with and without exercise intolerance
Change in coagulation biomarker - D-dimer | At diagnosis, 3 months and 12 months post-diagnosis
  Measure coagulation biomarker D-dimer (unit of measure: ng/mL) in participants with and without exercise intolerance
Change in coagulation biomarker - Thrombin generation | At diagnosis, 3 months and 12 months post-diagnosis
  Measure coagulation biomarker thrombin generation (unit of measure: nM·min) in participants with and without exercise intolerance
Change in coagulation biomarker - Fibrinolysis assay | At diagnosis, 3 months and 12 months post-diagnosis
  Measure coagulation biomarker fibrinolysis assay (unit of measure: % lysis) in participants with and without exercise intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Zia, MD, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (14):
- United States (14):
  - Arkansas Childrens Research Institute (ACRI), Little Rock, Arkansas
  - Johns Hopkins All Childrens Hospital, St. Petersburg, Florida
  - Emory University / Children's Heathcare Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Central Michigan University, Mount Pleasant, Michigan
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center / Children's Medical Center, Dallas, Texas
  - Cook Childrens Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: FUVID Website — http://www.utsouthwestern.edu/fuvid